CLINICAL TRIAL: NCT06634706
Title: Performance and Safety of Biology-Guided Radiotherapy Using the RefleXion Medical Radiotherapy System in in a Variety of Solid and Soft Tissue Tumors (BIOGUIDE-X2)
Brief Title: SCINTIX [BgRT} Using RMRS in Solid and Soft Tissue Tumors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RefleXion Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 985-00007
Record Dates: First submitted 2024-09-26; First posted 2024-10-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Thoracic Cancer; Head and Neck Cancer; Pelvic Cancer; Hepatobiliary Carcinoma in Situ; Retroperitoneal Cancer; Distributed and Orphan Tumors
MeSH Terms: conditions — Head and Neck Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 - Head and Neck Tumors (Other): Tumors in the following regions: Larynx, Salivary glands, Thyroid gland, Head and Neck lymph nodes, Oral cavity, Oropharynx, Nasopharynx, and Hypopharynx
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]
- Cohort 2 - Thoracic Tumors (Other): Tumors in the following regions: Thoracic lymph nodes, Thymus, Esophagus, and Breast,
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]
- Cohort 3 - Hepatobiliary Tumors (Other): Tumors in the following regions: Liver and intrahepatic ducts, Gallbladder, Extrahepatic bile ducts, and Hepatic lymph nodes,
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]
- Cohort 4 - Retroperitoneal Tumors & non-Hepatobiliary Abdominal Tumors (Other): Tumors in the following regions: Kidneys, Adrenal gland, Pancreas, Retroperitoneal lymph nodes, Stomach, Spleen, Small intestine, and Colon
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]
- Cohort 5 - Pelvic Tumors (Other): Tumors in the following regions: Prostate, Bladder, Ureter, Urethra, Cervix, Ovaries, Fallopian tubes, Vagina, Colon [Sigmoid], Rectum, Anus, and Pelvic lymph nodes.
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]
- Cohort 6 - Other and Orphan Tumors (Other): Tumors in the following regions: * Locations not listed in Cohorts 1-5, however; considered at physicians discretion i.e. Lymphoma [Head and Neck], Thorax, Abdomen, and Pelvis
  Interventions: Device: RefleXion X1 Radiotherapy System [Imaging Only]

INTERVENTIONS:
Device: RefleXion X1 Radiotherapy System [Imaging Only] — kVCT and FDG-PET imaging using the RefleXion X1 Radiotherapy System in different anatomical regions
  Other Names: RefleXion Medical Radiotherapy System

SUMMARY:
This study proposes 6 anatomic groupings which each can be defined similarly as the "head and neck" grouping above. These 6 groupings are: (1) Head and Neck, (2) Thoracic not including lung parenchymal, (3) Hepatobiliary and other non-hepatobiliary abdominal tumors, (4) Retroperitoneal, (5) Pelvic, and (6) Distributed or orphan. The study is designed to gather essential imaging data on the RefleXion Medical Radiotherapy System (RMRS) to validate the accuracy of FDG-directed BgRT, also known as SCINTIX therapy, in various anatomical groupings. Study subjects will go through the entire SCINTIX treatment workflow, including radiopharmaceutical administration and live PET imaging, but without turning on the treatment beam. Collected data will be used offline to generate the set of machine instructions that would have been used during treatment delivery to calculate the "emulated" BgRT dose distribution, i.e., what the delivered dose would have been had the treatment beam been turned on during the session. The 6th category ("Distributed or orphan") is meant to capture tumor types that can manifest across anatomies and/or for which utilization of stereotactic radiotherapy for treatment is relatively rare, with lymphomas being a prototypical example.

DETAILED DESCRIPTION:
Ablative radiotherapy has become an integral tool for the treatment of primary tumors and metastatic lesions across the human body. Because ablative radiotherapy techniques like stereotactic body radiotherapy (SBRT) and stereotactic radiosurgery (SRS) involve delivering high doses of radiotherapy in a few fractions, they have the potential to cause serious injury to normal tissues near the target lesion. Therefore, a standard concern for radiation oncologists is to conformally and precisely deliver ablative radiotherapy while maximally sparing surrounding organs and tissues. This goal is relevant throughout the anatomy and pertains as much to tumors in the head and neck as it does to those in the pelvis.

Biology-guided radiotherapy is a novel radiotherapy delivery mechanism that achieves precision by aiming beamlets of external radiotherapy by tracking PET emissions that originate from the target after it has taken up an injected radiotracer. Because the radiotherapy beamlets are guided to the tumor in real-time, this technology holds strong promise for reducing margins around the target and thereby reducing normal tissue toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 21 years.
2. A new or prior diagnosis of biopsy-proven cancer.
3. At least one active non-osseous primary or metastatic tumor that is located in one of the assigned anatomical groupings and dispositioned to undergo 3-5 fractions of SBRT. A lesion is considered active if viable malignancy is confirmed either by biopsy or by diagnostic imaging (as interpreted by the multidisciplinary care team).
4. Target tumor size ≥2cm and ≤5cm.
5. Target tumor is discrete and assessed by investigator to meet diagnostic PET screening criteria for BgRT candidacy:

   1. SUVmax≥6, as assessed on diagnostic PET/CT performed within 60 days of enrollment with no new intervening oncologic therapies.
   2. Ratio of target tumor SUVmax to SUVmean of local background region (defined as a 3 mm shell 1.5 cm from the target tumor) is greater than 6, as assessed on diagnostic PET/CT performed within 60 days of enrollment with no new intervening oncologic therapies.
6. ECOG Performance Status 0-3.
7. Must have completed any other oncologic therapies at least 15 days prior to planned start of study procedures (preferably 30 days) and must have no plans to initiate systemic therapy until after study follow up is complete -OR- must be recorded by physician to have an active lesion that is unresponsive to ongoing systemic therapy.
8. Females of childbearing potential should have a negative urine or serum pregnancy test within 14 days prior to initiation of study scans.

Exclusion Criteria:

1. Clinically significant blood glucose abnormalities that preclude a satisfactory FDG PET/CT scan.
2. Lung parenchymal and bone target tumors
3. At the physician's discretion regarding expected target motion, FDG-avid structures not intended for radiation are within:

   1. 3 cm from target on diagnostic PET/CT in directions where limited target motion is expected
   2. 4 cm from target on diagnostic PET/CT in directions where sizable target motion is expected
4. Known allergy to FDG.
5. Known psychiatric or substance abuse disorder that would interfere with conduct of the study.
6. Pregnant, breast-feeding or expecting to conceive during the study.
7. Patient weight exceeding the weight limit outlined per user manual.
8. Patients with pacemakers and other implantable devices deemed at high risk by the treating physician for complications secondary to radiotherapy, according to institutional guidelines and published guidelines (e.g. AAPM task group-203).
9. Active inflammatory bowel disease, scleroderma, or other disorder deemed by the treating physician to put the patient at risk for excess toxicity in the setting of external beam radiation therapy (EBRT) or FDG injection.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Emulated BgRT Delivery accuracy | Assessed for each emulated delivery through study completion, an average of 2 years
  The percent of radiotherapy fractions where the emulated BgRT dose distribution is shown to be consistent with the approved BgRT treatment plan (i.e., 95% of DVHDelivered points for the BTZ and OAR fall within bounded DVH of the approved BgRT plan).

SECONDARY OUTCOMES:
BgRT deliverability | Assessed for each emulated delivery through study completion,an average of 2 years
  Percent of fractions where there is concordance between physical and digital phantoms of emulated BgRT delivery derived from human subject PET emissions. Concordance is defined as a standard gamma index of 90% of pixels meeting the 3mm/3% deviation standard.

CONTACTS AND LOCATIONS:
Overall Officials: Sean S. Shirvani, MD, Study Director — RefleXion Medical Inc